CLINICAL TRIAL: NCT07294131
Title: Targeting Muscle Strength Loss Due to Hospitalization in Older Adults by Blood-flow Restriction Combined With an EMG-driven Serious Game
Brief Title: Targeting Muscle Strength Loss Due to Hospitalization in Older Adults by Blood-flow Restriction Combined With an Electromyography-driven Serious Game.
Acronym: GHOSTLY+
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Vrije Universiteit Brussel (Other)
Collaborators: Universitair Ziekenhuis Brussel (Other); University Hospital, Antwerp (Other); Universitaire Ziekenhuizen KU Leuven (Other); Universiteit Antwerpen (Other); KU Leuven (Other)
Responsible Party: Principal Investigator, Eva Swinnen, prof. dr., Vrije Universiteit Brussel
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CIV-25-06-053274; T000425N (Other Grant/Funding Number: Fonds Wetenschappelijk Onderzoek (FWO) Vlaanderen)
Record Dates: First submitted 2025-12-17; First posted 2025-12-19 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Hospital Associated Disability; Immobility; Older Adults (65 Years and Older)
Keywords: hospital-associated disability; HAD; muscle strength loss; blood flow restriction; BFR; serious games; EMG-driven rehabilitation; geriatric rehabilitation; older adults; lower-limb strength; non-weight-bearing; randomized controlled trial; RCT; physical deconditioning; hospitalization; electromyography; digital rehabilitation; implementation science; rehabilitation technology; exergaming; inpatient rehabilitation; strength training; GHOSTLY+
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: This is a multicenter, two-arm, parallel-group randomized controlled trial (RCT) using a Hybrid Type 1 effectiveness-implementation design.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Control Arm (Active Comparator): Participants in the control group will receive standard physiotherapy according to the usual clinical care procedures at the participating hospital site. No additional strength training, exercise tools, or exergaming interventions will be provided. Participants will be encouraged to remain active according to standard rehabilitation protocols but will not engage with the GHOSTLY+ system or any equivalent unsupervised strength training intervention.
  Interventions: Other: Standard Physiotherapy
- Intervention Arm (Experimental): Participants randomized to the intervention group will receive standard physiotherapy according to hospital protocol, supplemented with the GHOSTLY+ system.
  Interventions: Device: Gamified isometric strength training with blood flow restriction; Other: Standard Physiotherapy

INTERVENTIONS:
Device: Gamified isometric strength training with blood flow restriction — GHOSTLY+ is an interactive, EMG-driven serious game combined with blood flow restriction (BFR) therapy. Participants will undergo isometric quadriceps contractions guided by gameplay, with each session consisting of 3 sets of 12 contractions at 75% of their maximum voluntary contraction (MVC), as determined by in-app calibration. BFR will be applied using a smart cuff inflated to 50% of the participant's arterial occlusion pressure (AOP). Sessions will be performed independently by the patient during non-therapy time, with a minimum of 5 sessions per week over a 2-week period (or until discharge).
  Other Names: GHOSTLY+
  Arms: Intervention Arm
Other: Standard Physiotherapy — Usual standard-of-care physiotherapy as per hospital guidelines. This typically consists of supervised therapeutic sessions prescribed by the clinical team, including mobility exercises, transfer practice, and functional strengthening, depending on the patient's clinical needs and recovery stage. Participants do not perform structured lower-limb strength training outside of formal therapy sessions.
  Other Names: Standard Care

SUMMARY:
This study investigates a new training method designed to help older adults preserve their muscle strength during hospitalization. When older adults are admitted to the hospital and spend long periods in bed, their muscles can weaken very quickly. This condition is known as hospital-associated disability (HAD), and it can lead to longer hospital stays, reduced independence, and an increased risk of complications or even death. Conventional strength training with heavy weights is often too demanding or unsafe for frail patients, especially just after surgery or illness. As a safer alternative, this study combines light muscle exercises with a medically validated technique called blood flow restriction (BFR), which gently reduces blood flow to the leg to boost the effects of light exercises.

To make training more engaging and personalized, the GHOSTLY+ system was developed. This system consists of a game played on a tablet that responds to muscle activity through sensors placed on the skin. While playing, patients perform isometric muscle contractions (exercises where the muscles tighten without moving the joint) that help to maintain and rebuild strength. The system was carefully designed in collaboration with patients and therapists, and it has already been tested in a smaller pilot study at UZ Brussel.

The current study is a multicenter randomized controlled trial, taking place at UZ Brussel, UZ Antwerpen, and UZ Leuven. A total of 120 patients aged 65 or older will be recruited, all of whom are hospitalized and are unable to bear weight or transfer (e.g., from lying to seated position). Participants will be randomly assigned to one of two groups. One group receives standard physiotherapy. The other group receives standard therapy plus the GHOSTLY+ training program.

Those in the GHOSTLY+ group will train at least five times per week for two weeks, or until discharge from the hospital. Each training session lasts approximately 30 minutes and involves three sets of 12 muscle contractions, guided by the game. The difficulty is adapted to the individual's muscle strength, which is measured at the beginning of the training using a built-in calibration protocol. During the session, a smart cuff is applied to the upper leg to partially restrict blood flow - a technique shown to safely enhance muscle adaptation. The cuff is inflated to 50% of the individual's arterial occlusion pressure and deflated after the session ends. Before beginning, participants receive a short training session with a physiotherapist. Our pilot study (Debeuf et al., 2025) shows that most patients can use the system independently after about one hour of instruction.

Measurements and evaluations take place at three timepoints: before starting the training, after one week, and again at discharge. The main goal is to assess leg muscle strength, which will be measured using a handheld device called a dynamometer. In addition, researchers will collect information on:

* Muscle mass, via ultrasound of the thigh muscle
* Functional capacity, using a 30-second sit-to-stand test and a walking scale (Functional Ambulation Category)
* An index of independence in activities of daily living (Katz scale)
* Cognitive functioning, using the Mini-Mental State Examination (MMSE)
* Time spent bedridden and total length of hospital stay
* Therapy adherence and user experience, via usage data and questionnaires
* Muscle activity signals, such as fatigue, recorded during gameplay
* Implementation outcomes (collected via surveys, interview, site logbooks)

The study will also assess how easily the GHOSTLY+ system can be implemented in real hospital environments. This includes evaluations of user satisfaction, therapist feedback, and how consistently the system is used across hospital settings. Information will be gathered through structured interviews, surveys, and data logs from the app. These insights are crucial to understanding whether GHOSTLY+ can be broadly adopted in other hospitals in the future.

Blood flow restriction training is considered very safe when applied correctly and is already used in rehabilitation clinics and sports medicine worldwide. Over 300,000 sessions have been conducted internationally, with a very low rate of complications. Minor discomfort, such as temporary tightness or muscle fatigue, may occur, but the risk of serious side effects is extremely small.

By participating in this study, patients may benefit from improved muscle strength, reduced time spent in bed, and greater physical independence at discharge. The study also contributes to the development of more effective and enjoyable rehabilitation methods for older adults in hospitals.

DETAILED DESCRIPTION:
Hospitalization places older adults at significant risk for hospital-associated disability (HAD), a condition marked by a rapid and often severe decline in muscle strength and function due to immobility. Research has shown that adults aged 65 and older can lose up to 15% of their lower-limb strength within a single week of bed rest, and as much as 5% of muscle mass per day. These declines not only prolong the length of hospital stay but also increase dependence, impair mobility, and elevate the risk of mortality. While high-load resistance training is considered the gold standard for preventing muscle loss, it is often contraindicated or simply unfeasible for frail or post-surgical patients. This creates an urgent need for effective, low-impact alternatives to preserve physical function during hospitalization.

Blood flow restriction (BFR) training has emerged as one such alternative. It works by partially occluding arterial blood flow and fully restricting venous return in a limb using a pressure cuff, thereby enhancing the effects of low-load exercise. BFR has been demonstrated to stimulate muscle hypertrophy and strength gains in various populations, including older adults, and has been shown to be safe in over 300,000 reported clinical sessions. In addition to physical limitations, another major challenge in hospital rehabilitation is poor adherence. Many patients fail to complete unsupervised therapy exercises, largely due to low motivation. Serious games - interactive applications designed with a therapeutic goal - have shown promise in improving engagement, but most are not designed specifically for clinical use or individualized for the needs of hospitalized older adults.

To address these challenges, the GHOSTLY+ system was developed. GHOSTLY+ is a mobile rehabilitation solution combining gamified muscle training with BFR, designed to be used during non-therapy time in hospitalized older adults. The system is based on a serious game app that transforms muscle contractions, measured via surface electromyography (EMG), into in-game actions. By engaging patients in a playful yet physiologically grounded environment, the system aims to increase motivation and ensure proper exercise intensity, even without the use of weights or active movement. GHOSTLY+ includes automated difficulty adjustment based on real-time EMG input and follows evidence-based parameters for strength training: isometric contractions at approximately 75% of each patient's maximum voluntary contraction (MVC), performed three times per session with 12 repetitions each set.

The clinical study described here is a multicenter, randomized controlled trial (RCT) using a Hybrid Type 1 design. The trial will be conducted at three hospitals in Belgium (UZ Brussel, UZ Antwerpen, and UZ Leuven) and will enroll 120 older adults aged 65 years or above who are hospitalized, unable to bear weight or transfer independently, are expected to remain hospitalized for approximately 14 days, and are at high risk of muscle strength loss due to prolonged immobility. Participants will be randomly assigned to one of two groups. The control group will receive standard physiotherapy as prescribed in the hospital. The intervention group will receive standard care supplemented with the GHOSTLY+ system. Participants will use GHOSTLY+ for at least five sessions per week, over two weeks or until discharge, depending on their hospital stay duration.

Each GHOSTLY+ session begins with the application of a smart BFR cuff to the upper thigh of the target leg. The cuff automatically measures the arterial occlusion pressure (AOP) and inflates to 50% of this value, a level known to be effective while minimizing discomfort. Participants are then guided through an in-app calibration process in which they perform three maximal isometric contractions. Based on these readings, the system determines the individual's MVC and sets the game difficulty to 75% of that value. During gameplay, patients must complete three levels per session, with each level representing a set of twelve muscle contractions. Rest periods of two minutes are provided between sets. Based on a previous proof-of-concept study conducted at UZ Brussel (Debeuf et al., 2025), most patients are able to use the system independently after one hour of training. Physiotherapists at each site will be trained to guide this initial setup until patients are independently capable of setting up the GHOSTLY+ system.

The primary outcome of this study is lower-limb muscle strength at hospital discharge, assessed using a handheld MicroFet dynamometer. Secondary outcomes include muscle mass measured via ultrasound imaging of the rectus femoris, functional performance assessed through the 30-second sit-to-stand test and the Functional Ambulation Category, independence in activities of daily living using the Katz scale, time spent bedridden, total length of hospital stay, and patient-reported outcomes related to satisfaction and usability of the intervention. Cognitive status will be assessed using the Mini-Mental State Examination (MMSE), and additional analysis will be performed on EMG data to extract neuromuscular parameters such as signal amplitude and fatigue index. In addition to clinical and physiological data, patients and therapists will participate in implementation data collection via surveys, interviews, and site logbooks, in line with the Consolidated Framework for Implementation Research (CFIR).

Data will be collected at three time points: before the intervention (baseline), at the end of the first week, at the end of two weeks, or at hospital discharge if earlier. Randomization will be performed using a web-based system, with assessors blinded to group allocation to reduce bias. Participants will receive a study-specific ID and will be instructed not to disclose their group assignment to those collecting outcome measures.

Beyond evaluating clinical efficacy, the trial incorporates a robust implementation evaluation. Using the Consolidated Framework for Implementation Research (CFIR) and Proctor's framework, the study will examine key real-world indicators such as acceptability, adoption, fidelity, feasibility, penetration, and sustainability. Data will be gathered through staff surveys, administrative records, structured interviews, app usage data, and focus groups with healthcare professionals and patients. The qualitative data will be analyzed using content analysis and reflexive thematic analysis to identify implementation facilitators and barriers.

The study is powered to detect a 15% difference in lower-limb strength preservation between the intervention and control groups. Analysis will include repeated measures ANOVA, regression modeling, and subgroup analysis to explore the impact of baseline mobility status or cognitive performance. All data will be monitored for quality and completeness, and any serious adverse events will be reported to the competent authorities following the applicable safety guidance under the EU Medical Device Regulation.

Following trial completion, the research team will prepare an implementation package, including an e-learning training module for clinical staff, a Grol & Wensing-based implementation guideline, and a business case for broader adoption. Results will be disseminated through academic publications, clinician workshops, hospital presentations, and patient information campaigns.

In summary, this trial evaluates GHOSTLY+, a novel rehabilitation system combining blood flow restriction and EMG-guided gamified strength training for hospitalized older adults. It is designed to preserve muscle strength, reduce physical decline during bedrest, and boost adherence to therapy using interactive digital technology. By embedding implementation science into its structure, the study aims to not only prove the effectiveness of GHOSTLY+ but also support its sustainable integration into routine hospital care.

ELIGIBILITY:
PATIENTS

Inclusion Criteria:

* Hospitalized, and expected to remain hospitalized for approximately 14 days
* 65+ yrs
* Unable to bear weight or transfer independently and at high risk of muscle strength loss due to prolonged immobility

Exclusion Criteria:

* Contraindications for physical exercise as assessed by the treating physician using the risk assessment tool proposed by Kacin et al. (2015) (can be overruled by the physician)
* Contraindications for blood flow restriction as assessed by the treating physician (can be overruled by the physician)
* Cognitive impairment (MMSE score < 19)
* Any condition that renders the patient unable to understand instructions or safely interact with the GHOSTLY+ system

THERAPISTS

Inclusion Criteria:

Therapists will be included if

* They are licensed physiotherapists employed at one of the three participating clinical sites
* They are involved in the daily rehabilitation of hospitalized older adults.

Exclusion Criteria:

Therapists will be excluded from participation if

* They are unable or unwilling to complete the GHOSTLY+ training
* They are not directly involved in the care of eligible patients during the study period
* They express any conflict of interest or ethical concern that may compromise the integrity of the study

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2029-01-01 (Estimated); Study Completion 2029-01-01 (Estimated)

PRIMARY OUTCOMES:
Maximal isometric muscle strength | From enrollment to the end of treatment at 2 weeks (or until hospital discharge if earlier).
  Maximal isometric muscle strength of the lower limbs will be assessed using a handheld dynamometer (MicroFET or equivalent). The test involves measuring the peak isometric force generated by the quadriceps muscle group during a voluntary contraction against resistance, while the participant is in a standardized seated position. Each participant will perform three maximal voluntary contractions (MVCs) with sufficient rest between trials. The highest recorded peak force (Newtons) will be used as the representative value. Testing will be conducted at three time points: baseline (T0), after one week (T1), and at two weeks or at the time of hospital discharge, whichever occurs first (T2). Outcome assessors are blinded to group allocation. The change in maximal isometric quadriceps strength (Newtons) from baseline to discharge will serve as the primary endpoint to evaluate the intervention's effectiveness in preserving muscle strength during hospitalization.

SECONDARY OUTCOMES:
Electromyography (EMG) Signal Analysis | At the end of week 1, and the end of treatment at 2 weeks (or until hospital discharge if earlier).
  Analyses will be performed on EMG data to extract the neuromuscular parameter: signal amplitude.
Cross-sectional area of the Rectus Femoris Muscle | From enrollment to the end of treatment at 2 weeks (or until hospital discharge if earlier).
  The muscle mass of the m. rectus femoris will be assessed using a bedside ultrasound system. The cross-sectional area (CSA) of the muscle will be measured in a supine position at a standardized mid-thigh location. Assessments will occur at baseline (T0), week 1 (T1), and discharge (T2). This outcome is intended to capture muscle architecture changes associated with strength loss or preservation.
Functional performance - 30 second sit-to-stand test | From enrollment to the end of treatment at 2 weeks (or until hospital discharge if earlier).
  If medically permitted (i.e., participant is weight-bearing), functional lower-limb endurance will be measured using the 30-second sit-to-stand test (30s-STS). Participants will be asked to rise from a standardized chair to a full standing position and sit back down as many times as possible in 30 seconds. Standardized instructions and encouragement will be used. This test is a validated measure of functional strength and endurance. Performance will be assessed at T0, T1, and T2.
Functional ambulation category (FAC) | From enrollment to the end of treatment at 2 weeks (or until hospital discharge if earlier).
  The Functional Ambulation Category (FAC) is a 6-point scale used to assess the level of independence in walking. It ranges from 0 (non-functional ambulation) to 5 (independent ambulation in all environments). Assessment is performed at T0, T1 and T2. FAC will help determine the extent to which patients regain or retain ambulatory capacity during hospitalization.
Time spent bed- or chair-ridden | From enrollment to the end of treatment at 2 weeks (or until hospital discharge if earlier).
  The cumulative number of hours spent bed- or chair-ridden during the hospital stay will be recorded at T2, using daily nursing records and physiotherapy logs. This outcome serves as an indicator of mobility and physical activity during hospitalization.
Hospital length of stay | From enrollment to the end of treatment at 2 weeks (or until hospital discharge if earlier).
  The total length of hospital stay, from admission to discharge, will be extracted from hospital records at T2. This metric will help determine whether the intervention has an effect on overall hospitalization duration, potentially through earlier recovery or functional independence.
Adherence: number of sessions | From enrollment to the end of treatment at 2 weeks (or until hospital discharge if earlier).
  Adherence to the intervention will be tracked automatically through usage logs embedded in the GHOSTLY+ software, and will be extracted at T1 and T2. Metric 1: number of sessions completed.
Adherence: duration of play | From enrollment to the end of treatment at 2 weeks (or until hospital discharge if earlier).
  Adherence to the intervention will be tracked automatically through usage logs embedded in the GHOSTLY+ software, and will be extracted at T1 and T2. Metric 2: duration of play per session.
Adherence: percentage of completed repetitions | From enrollment to the end of treatment at 2 weeks (or until hospital discharge if earlier).
  Adherence to the intervention will be tracked automatically through usage logs embedded in the GHOSTLY+ software, and will be extracted at T1 and T2. Metric 3: percentage of completed repetitions (%).
Usability and satisfaction | From enrollment to the end of treatment at 2 weeks (or until hospital discharge if earlier).
  Patient-reported usability and satisfaction with the GHOSTLY+ system will be measured using customized questionnaires developed for this study. It will assess ease of use, clarity of instructions, perceived benefit, and overall satisfaction using Likert-scale questions. Administered at discharge (T2), the goal is to evaluate patient experience and barriers/facilitators for future implementation.
Katz Index of Independence in Activities of Daily Living | At enrollment, and at the end of treatment at 2 weeks (or until hospital discharge if earlier).
  The purpose of the Index of ADL, or Katz ADL, is to monitor the prognosis and treatment of older adults and chronically ill individuals. In particular, the Katz ADL measures a person's independence in common activities of daily living (ADL).
EQ-5D QOL | At enrollment, and at the end of treatment at 2 weeks (or until hospital discharge if earlier).
  The EQ-5D is a standardized instrument for measuring health-related quality of life (QoL), consisting of five dimensions: mobility, self-care, activities of daily living, pain/discomfort, and anxiety/depression. It consists of a descriptive system and a visual analog scale (EQ VAS).
Charlson Comorbidities Index | At enrollment.
  The Charlson Comorbidity Index predicts the mortality for a patient who may have a range of concurrent conditions (considering a total of 17 categories). A score of zero means that no comorbidities were found; the higher the score, the higher the predicted mortality rate and the lower the predicted ten-year survival.
Mini Mental State Examination | At enrollment.
  The Mini-Mental State Examination (MMSE) is a brief, 11-question test used to screen for cognitive impairment by assessing a person's orientation, attention, memory, language, and visual-spatial skills.
Usefulness, Satisfaction, and Ease of Use (USE) | At 2 weeks (or until hospital discharge if earlier).
  The Usefulness, Satisfaction, and Ease of Use (USE) questionnaire is a validated 30-item scale designed to assess users' perceived usefulness, satisfaction, and ease of use of a system. Scores reflect how well the system supports task performance, how pleasant it is to use, and how intuitively users can interact with it.
System Usability Scale (SUS) | At 2 weeks (or until hospital discharge if earlier).
  The System Usability Scale (SUS) is a widely used 10-item questionnaire that provides a global measure of perceived system usability.Higher scores indicate better usability.

OTHER OUTCOMES:
Implementation Outcome: Acceptability | From the start of the study until maximally one year later.
  Acceptability refers to how suitable, satisfying, or agreeable the GHOSTLY+ intervention is perceived to be by its users - including both patients and healthcare providers. This will be assessed through structured surveys and semi-structured interviews or focus groups conducted after the intervention period. Topics will include perceptions of usefulness, ease of use, clarity of instructions, and perceived value. Data will be analyzed qualitatively using thematic analysis and quantitatively via survey responses to gauge overall user satisfaction and alignment with clinical needs.
Implementation Outcome: Adoption | From the start of the study until maximally one year later.
  Adoption reflects the initial decision and action to try or employ the GHOSTLY+ system by healthcare professionals at each participating hospital site. This will be measured using administrative logs, recruitment records, and surveys documenting how many physiotherapists or staff chose to engage with the intervention, and what factors influenced their willingness to do so. Qualitative interviews will further explore facilitators and barriers influencing the uptake of the system in routine clinical workflows.
Implementation Outcome: Fidelity | From the start of the study until maximally one year later.
  Fidelity refers to the degree to which the GHOSTLY+ intervention was delivered as intended. This includes adherence to the planned session structure (e.g., 3 sets of 12 repetitions at 75% MVC with BFR), use of app features such as calibration and real-time feedback, and proper application of the BFR cuffs. Fidelity will be monitored via usage logs, therapist checklists, and adherence data from app dashboards. Deviations from the protocol will be documented and analyzed to understand variability in delivery and potential impact on outcomes.
Implementation Outcome: Feasibility | From the start of the study until maximally one year later.
  Feasibility captures the extent to which GHOSTLY+ can be successfully used in a real-world clinical setting, given practical constraints such as staffing, time, space, and technology integration. It will be assessed through clinician and staff surveys, logbooks, and feedback interviews. Indicators include training burden, technical difficulties, workflow fit, and perceived logistical challenges.
Implementation Outcome: Penetration | From the start of the study until maximally one year later.
  Penetration refers to the degree of integration of GHOSTLY+ into the existing infrastructure at each hospital site during the study. This includes how deeply the intervention is embedded in routine care, how many eligible patients received the intervention, and how widespread its use was among trained therapists. Data will come from administrative logs, therapist reports, and app usage metrics, complemented by qualitative exploration of contextual factors affecting implementation depth.
Implementation Outcome: Sustainability | From the start of the study until maximally two years later.
  Sustainability assesses the extent to which the GHOSTLY+ intervention is maintained or likely to be maintained in clinical practice beyond the trial period. It includes both individual-level (e.g., staff willingness to continue use) and organizational-level (e.g., hospital policies, resource allocation) factors. Data will be collected through follow-up interviews with site leads and therapists, focused on intentions for long-term use, perceived value, and infrastructure readiness.

CONTACTS AND LOCATIONS:
Overall Officials: Eva Swinnen, prof. dr., Principal Investigator — Vrije Universiteit Brussel
Locations (3):
- Belgium (3):
  - Universitair Ziekenhuis Antwerpen, Antwerp
  - Universitair Ziekenhuis Brussel, Brussels
  - Universitair Ziekenhuis Leuven, Leuven

IPD SHARING:
Plan to Share IPD: Undecided